CLINICAL TRIAL: NCT02522845
Title: Multicentre Randomised Controlled Trial of Compression Therapy Following Endothermal Ablation (COMETA)
Brief Title: Compression Therapy Following Endothermal Ablation
Acronym: COMETA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15/LO/0181
Record Dates: First submitted 2015-08-04; First posted 2015-08-13 (Estimated); Results first posted 2020-07-27 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-08

CONDITIONS: Varicose Veins
Keywords: Varicose Veins; Compression Stockings; Laser Ablation; Catheter Ablation, Radiofrequency
MeSH Terms: conditions — Varicose Veins

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Compression (Active Comparator): Patients randomised to this group will be asked to wear Class II compression stockings for 1 week
  Interventions: Device: Class II Compression Stockings (no specific device used)
- No Compression (No Intervention): Patients randomised to this group will not be provided with any compression

INTERVENTIONS:
Device: Class II Compression Stockings (no specific device used) — This study will be looking at the effect of compression therapy in patients having endothermal treatment for truncal incompetence of their varicose veins
  Arms: Compression

SUMMARY:
This study will be looking at the effect of compression therapy in patients having endovenous treatment for truncal incompetence of their varicose veins using either radiofrequency ablation (RFA) or endovenous laser therapy (EVLT). Patients will be randomised to either the compression group (group A) or the no compression group (group B).

The pain scores, compliance, quality of life scores, occlusion rate at 6 months as well as the cost effectiveness of each intervention will be assessed.

DETAILED DESCRIPTION:
Background

Varicose veins are common and are known to affect approximately one third of the population. Chronic venous disease (CVD) has been shown to have a negative impact on the quality of life of patients and treatment of varicose veins has been demonstrated to lead to improvement in the quality of life of patients. Over the past decade, new endovenous techniques have been introduced and these are felt to be cost-effective, especially, when performed in an outpatient or 'office-based' setting.

There is currently uncertainty about the use of compression stockings following treatment of varicose veins. In their consensus statement in 2008, the International Union of Phlebology (IUP) stated that there is good evidence for using compression in certain clinical indications. These include the management of telangiectasia after sclerotherapy, varicose veins in pregnancy, prevention of thromboembolism and healing of ulcers. However, a few questions remain unanswered, such as the length of treatment and level of compression to be used6. The Society for Vascular Surgery and the American Venous Forum recommend using compression stockings post-operatively for 1 week to prevent haematoma formation, pain and swelling. The 2013 NICE Guidelines on Varicose Veins in the Legs recommended the use of compression hosiery for no more than 7 days after interventional treatment for varicose veins. However, due to current uncertainty of compression bandaging or hosiery compared to no compression after interventional treatment for varicose veins, the NICE Guideline Development Group have advocated further research to evaluate the clinical and cost effectiveness of this post-procedure intervention. The guidelines also suggested looking into the length of time compression bandaging should be worn if it shown to be beneficial.

Several researchers have looked into the practice of using compression after venous ablation. In a survey of the management of varicose veins by the members of the Vascular Society of Great Britain and Ireland, Edwards et al. found that the majority of surgeons used bandages post-operatively, with 49% using elastic bandages. The literature on the use of compression stockings following treatment of varicose vein is limited.

Between December 2006 and February 2008, Bakker and colleagues conducted a prospective randomised controlled trial on the use of compression stockings after endovenous laser ablation of the great saphenous vein. One hundred and nine patients were approached with 93 finally randomised to use compression stockings for 2 days (Group A) and 7 days (Group B), respectively. All patients were followed up for 3 months post-treatment and the visual analogue scale (VAS) for pain was recorded at 48 hours, 1 week and 6 weeks. A physical examination and quality of life was assessed at 1 week and 6 weeks. Occlusion rate at the 3 month point was also evaluated. Physical function and vitality was shown to be significantly better in group B at 1 week follow-up, but there was no statistically significant difference at 6 weeks. At 1 week, it was also noted that the VAS score in group B (VAS score 2.0 ± 1.1) was significantly lower than in patients wearing compression stockings for 48 hours (VAS score 3.7 ± 2.1) (p≤0.001)10. No significant difference was, however, observed at 6 weeks post-procedure. Limitations of the study include the high drop out of the trial (40 out of the initial 109 approached) and the absence of any phlebectomies or sclerotherapy in the patients.

Elderman et al. carried out a randomised trial to assess the effect of compression stockings after endovenous laser therapy (EVLT) for great saphenous vein incompetence. Patients' reported pain scores and quality of life scores was evaluated on the day of the procedure, 2-3 days afterwards and 2-6 weeks post-procedure. A total of 111 patients were randomised to stockings (n=55) and no stockings (n=56). There was a statistically significant difference in the pain scores in favour of the stockings group up to day 7, but this difference was no longer present by week 6. There was also a greater use of analgesia in patients in the no stockings group compared to patients wearing stockings (p<0.05). In addition, patients wearing stockings reported a statistically significantly higher score of satisfaction at 2 days (4.44 vs 4.15) and at 6 weeks (4.59 vs 4.18). The absolute difference was, however, small. Two notable limitations of the study were the high level of drop outs (16 from each group) and the absence of any blinding.

Hamel-Desnos et al. undertook a randomised controlled trial looking at the effect of compression in patients receiving foam sclerotherapy of the saphenous vein. They noted that patients with compression had similar pain and quality of life scores to patients not wearing any compression. They concluded that additional use of compression had no impact on the effectiveness of obliteration of veins, satisfaction scores, symptoms and quality of life, and that further controlled trials was needed to answer the question of whether using compression results in any difference to the outcome of varicose vein procedures.

The investigators, therefore, propose to undertake a multicentre randomised study looking at the effect of compression therapy after endovenous thermal ablation.

Description

This will be a multicentre randomised clinical trial looking at the impact of wearing or not wearing compression stocking following endothermal ablation (either endovenous laser treatment (EVLT) or radiofrequency ablation (RFA)) of incompetent truncal veins. Those requiring concurrent phlebectomies or foam injection will be excluded.

Patients will be randomised into group A (compression) and group B (no compression). Only the use of compression will be randomised while the decision as to which treatment to use will be at the discretion of the clinical team.

Target Population

Patients referred for treatment of symptomatic varicose veins will be recruited if they are found to have primary great saphenous (GSV) or small saphenous vein (SSV) incompetence on colour duplex scan.

Intervention

Patients will be randomised to have compression (group A) or no compression (group B). The compression therapy used will be Class II compression stockings. The treatment offered will be endothermal ablation (either endovenous laser treatment (EVLT) or radiofrequency ablation (RFA)) of incompetent truncal veins. Concurrent phlebectomy or foam sclerotherapy will not be carried out.

Patients randomised to group A will be asked to wear compression stockings for 1 week.

Patients randomised to group B will not be provided with any compression.

At baseline, patients will be asked to fill quality of life questionnaires (EQ-5D, AVVQ and CIVIQ) and will have their clinical scores assessed (CEAP and VCSS). On discharge after their varicose vein intervention, they will then be provided with a diary to record their post-procedural pain every day for 10 days using a validated visual analogue scale (VAS) as well as to record when they return to their normal activities and are back to work. They will also be asked to attend a follow-up in 2 weeks and at 6 months.

Patients' GP will also be sent a letter to inform them of their patient's participation in the study.

Follow-up

Patients will be followed up in the outpatient clinic at 2 weeks and 6 months.

Follow-up at 2 Weeks At the 2 weeks' follow-up, the diary containing details of the pain scores and how soon patients were able to return to normal activities/work will be collected. In addition, patients will be asked about any bruising or phlebitis they have had in the two weeks after their procedure and how compliant they have been with the compression. They will be examined and the Venous Clinical Severity Score (VCSS) will be recorded. They will also be asked to fill in the EQ-5D, AVVQ and CIVIQ scores.

Follow-up at 6 Months At the 6 months follow-up, patients will be examined and their VCSS will be recorded. They will also be asked to fill the EQ-5D, AVVQ and the CIVIQ scores. They will have a venous Duplex scan to determine occlusion of the treated vein.

Sample Size and Study Duration

The study team estimated the sample size needed to observe a difference of at least 10mm in the VAS score, with a standard deviation of 20mm. With power at 80% and 5% significance equivalence, the study would need to recruit 128 patients (64 per group) to show a difference.

Previous studies looking at compression stockings have shown drop out rates close to 37% at 3 months10. Therefore, if an estimated drop out rate of about 40% by 6 months is used, at least 214 patients would need to be recruited. If at least 2 patients per week are recruited, this will be approximately a total of 208 patients that could potentially be randomised over the course of two years.

With 6 months follow-up, therefore, the study will be running for 24 months with a target recruitment of 214 patients.

Settings The study will be conducted at the Imperial College NHS Trust

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years of age
* Symptomatic GSV or SSV vein reflux > 0.5 seconds on colour Duplex

Exclusion Criteria:

* Current DVT
* Recurrent varicose veins
* Patients requiring adjuvant treatment of varicose veins
* Arterial disease (ABPI<0.8)
* Vein diameter < 3mm
* Patient who are unwilling to participate
* Inability or unwillingness to complete questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Charing Cross Hospital, Imperial College London, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial period ran from May 2015 to December 2018
Pre-assignment Details: Patients not meeting inclusion criteria
Groups:
- Compression: Patients randomised to this group will be asked to wear Class II compression stockings for 1 week after 24 hours of compression bandaging
  Class II Compression Stockings (no specific device used): This study will be looking at the effect of compression therapy in patients having endothermal treatment for truncal incompetence of their varicose veins
- No Compression: Patients randomised to this group will not be provided with any compression after 24 hours of compression bandaging
Period: Overall Study
Arm/Group | Compression | No Compression
Started | 100 | 104
Completed | 63 | 69
Not Completed | 37 | 35

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Compression | No Compression | Total
Number analyzed (Participants) | 100 | 104 | 204
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.7 (17) | 49.6 (15) | 49.7 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 58 | 100
  Male | 58 | 46 | 104
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 100 | 104 | 204
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 27.3 (5) | 27.0 (7) | 27.1 (6)

OUTCOME MEASURES:

1. Primary Outcome: Patient's Post-procedure Pain Score Using a Visual Analogue Scale (VAS)
Description: Patients indicating level of pain they were having using a VAS scale. The scale is a 100mm line drawn going from 0-100 (0=no pain; 100=worse pain)
Time Frame: Up to 10 days
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | Compression | No Compression
Number analyzed (Participants) | 63 | 69
mm | 18.7 [7.58 to 36.9] | 27.8 [13.0 to 53.6]

2. Secondary Outcome: The Generic Quality of Life Score Using the EQ-5D Score
Description: The EQ-5D is a quality of life scale with 5 statements with 3 possible answers. Each answer is scored from 1 to 3 (1=best; 3=worse). Each answer is then collated (from 11111 to 33333). Using a calculator, these answers are translated into a scale which goes from -0.073 to 1.0 (-0.073= worse; 1=best).
Time Frame: Up to 6 months
Population: This is a patient-completed scoring instrument and not every patient filled/completed this.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Compression | No Compression
Number analyzed (Participants) | 46 | 44
units on a scale | 0.761 [0.690 to 1.0] | 0.891 [0.722 to 1.0]

3. Secondary Outcome: The Specific Quality of Life Score Using the Aberdeen Varicose Vein Questionnaire (AVVQ) Score
Description: The disease-specific AVVQ score has 13 items with different scoring for each item. The final scores are added and then the percentage is calculated. The final score goes from 0 to 100 (0=best; 100= worse)
Time Frame: Up to 6 months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Compression | No Compression
Number analyzed (Participants) | 46 | 44
units on a scale | 7.3 [3.0 to 16.3] | 10.1 [2.5 to 16.7]

4. Secondary Outcome: The Specific Quality of Life Score Using the CIVIQ Score
Description: This is a quality of life scale going from 0 to 100 (0=best; 100=worse)
Time Frame: Up to 6 months
Population: This is a patient-completed scoring instrument and not every patient filled/completed this.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Compression | No Compression
Number analyzed (Participants) | 46 | 44
units on a scale | 7.1 [1.8 to 20.5] | 5.4 [1.8 to 16.1]

5. Secondary Outcome: The Clinical Score Using the Venous Clinical Severity Score
Description: This is a scoring system with 10 items graded from 0 to 3 (0=best/absent; 3=worse/present). The individual scores are then added to obtain the final score (0=best; 30=worse).
Time Frame: Up to 6 months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Compression | No Compression
Number analyzed (Participants) | 46 | 44
units on a scale | 2 [1.0 to 4.0] | 1 [1 to 3]

6. Secondary Outcome: The Degree of Bruising and Phlebitis
Description: The degree of bruising and phlebitis will be assessed using a pre-determined score (0=0%; 1= <25% of treated vein affected; 2 = 25-50% ; 3 = 50-75%; 4 = 75-100% and 5 = extending beyond the treated vein. Using this pre-defined score, patients were divided into two groups (those with a score of 1 or less, and those with a score of 2-5).
  The outcome measure is the percentage of patients with a score of 1 or less.
Time Frame: Up to 6 months
Measure: Number; unit: percentage
Arm/Group | Compression | No Compression
Number analyzed (Participants) | 63 | 69
percentage | 85 | 80

7. Secondary Outcome: The Number of Days After Treatment That Patients Were Compliant With the Intervention
Description: This looked at the number of days since intervention that patients stopped wearing compression stockings if they were allocated to the compression group
Time Frame: Up to 3 weeks
Population: Patient in no compression group not provided with stockings
Measure: Median (Full Range); unit: day
Arm/Group | Compression | No Compression
Number analyzed (Participants) | 100 | 0
day | 7 [0 to 20] |

8. Secondary Outcome: The Time Taken to Return to Work and Normal Activities
Description: This looked at the number of days since intervention before patients are able to resume their normal activities or go back to work
Time Frame: 1 month
Measure: Median (Inter-Quartile Range); unit: day
Arm/Group | Compression | No Compression
Number analyzed (Participants) | 63 | 69
day | 2 [1 to 3] | 3 [2 to 4]

9. Secondary Outcome: Occlusion Rates at 6 Months
Description: This looked at the occlusion of the target vein following treatment as assessed by an ultrasound duplex
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Compression | No Compression
Number analyzed (Participants) | 46 | 44
Participants | 41 | 41

10. Secondary Outcome: The Cost of the Intervention
Description: This looks at the cost of both interventions
Time Frame: 1 week
Reporting Status: Not Posted, anticipated posting 2023-12

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Compression | No Compression
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/104
Serious Adverse Events (participants affected / at risk) | 0/100 | 1/104
Other Adverse Events (participants affected / at risk) | 15/100 | 21/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Compression (N=100) | No Compression (N=104)
DVT (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Compression (N=100) | No Compression (N=104)
Superficial Vein Thrombosis (SVT) (Vascular disorders) | 0 (0) | 0 (0) — SVT (also referred as thrombophlebitis) is thombosis within the superficial veins
Ecchymosis (Vascular disorders) | 15 (15) | 21 (21) — Bruising arising from treatment

LIMITATIONS AND CAVEATS:
1. Power of the study was decreased from 90% to 80%.
2. The use of analgesia was not recorded so that it is unclear whether the pain score observed was with or without analgesia.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-19): https://cdn.clinicaltrials.gov/large-docs/45/NCT02522845/Prot_SAP_000.pdf